CLINICAL TRIAL: NCT07369154
Title: A 52 Week, Open Label Safety and Tolerability Study of LB-102 in Adult Patients With Schizophrenia
Brief Title: 52-week Open Label Safety-Tolerability Study
Acronym: NOVA3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: LB Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB-102-010
Record Dates: First submitted 2025-12-26; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LB-102 (Other): An open label study
  Interventions: Drug: LB-102

INTERVENTIONS:
Drug: LB-102 — LB-102 flexible dosing 50 mg - 100 mg

SUMMARY:
Phase 3, open label, multicenter study designed to assess the long term safety and tolerability of LB-102 for the treatment of adult patients with stable schizophrenia

DETAILED DESCRIPTION:
Phase 3, open label, multicenter study designed to assess the long term safety and tolerability of LB-102 for the treatment of adult patients with stable schizophrenia who are experiencing inadequate response or who are having issues with side effects, general tolerability, or overall effectiveness of their current antipsychotic medication and desire to change medications, or who have completed their participation in current LB-102 clinical studies

ELIGIBILITY:
Inclusion Criteria:

* Provide ICF
* Patients clinically stable PANSS </= 70 at screening
* CGI-S </+ 3 at screening
* Medically stable
* BMI 18 -40
* Taking oral antipsychotic treatment for at least 30 days
* Have stable living environment

Exclusion Criteria:

* Sexually active M/F patients not willing to use highly effective contraception
* Breast feeding
* History of treatment resistance to schizophrenia medications
* DSM-5 current diagnosis other than schizophrenia
* Risk of suicidal behavior
* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate long term safety and tolerability of LB-102 by evaluating the number of adverse event, incidence of treatment emergent events. | 52 weeks
  Overall adverse events, serious adverse events, incidence of treatment emergent events and adverse events which lead to study discontinuation

SECONDARY OUTCOMES:
Evaluate long term safety and tolerability | 52 weeks
  Evaluating the safety of treatment by number of adverse events
Evaluate long term safety and tolerability | 52 weeks
  Evaluating the safety of treatment by change in vital signs, electrocardiogram (QTC), and weight/height for BMI
Evaluate long term safety and tolerability | 52 weeks
  Evaluating the safety of treatment by conducting physical examinations
Assess the long-term effectiveness determined by Positive and Negative Syndrome Scale (PANSS) | 52 weeks
  Change in Positive and Negative Syndrome Scale (PANSS) from Baseline to end of treatment where a decrease in score likely indicate response to treatment whereas an increase in score may indicate a worsening of disease where an increase in the scale score may indicate a worsening of disease and decrease in score likely indicates response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John Kane, MD, Principal Investigator — Northwell Health

IPD SHARING:
Plan to Share IPD: No